CLINICAL TRIAL: NCT00126243
Title: Multicenter, Open Label, Phase II Trial to Evaluate the Efficacy and Safety of Treatment With Rituximab + CHOP Regimen in Patients With HIV Related Non-Hodgkin's Lymphomas. ANRS 085 Rituximab
Brief Title: Efficacy of Rituximab and Cyclophosphamide, Doxorubicin, Vincristine, Prednisone (CHOP) in Patients With HIV Associated Non-Hodgkin's Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Collaborators: Hoffmann-La Roche (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANRS 085 Rituximab
Record Dates: First submitted 2005-08-02; First posted 2005-08-03 (Estimated); Last update posted 2005-08-17 (Estimated); Status verified 2005-08

CONDITIONS: AIDS Related Lymphoma
Keywords: AIDS related Lymphoma; chemotherapy; rituximab
MeSH Terms: conditions — Lymphoma, AIDS-Related | interventions — Rituximab

INTERVENTIONS:
Drug: rituximab
Drug: CHOP

SUMMARY:
Most treatment procedures in AIDS-related lymphomas disclose a relatively poor outcome for patients with low response rates, high number of relapses and AIDS events. The addition of rituximab to the standard regimen - CHOP could improve the outcome of these patients. The aim of the trial is to evaluate the safety and efficacy of rituximab when added to the CHOP regimen in patients with newly diagnosed AIDS-related non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
HIV infection is associated with a high incidence of AIDS-related lymphomas (ARL). Since the use of highly active antiretroviral therapy (HAART), the incidence of AIDS-defining illnesses has decreased, leading to a significant improvement in survival of HIV-infected patients. The incidence of ARL has decreased in a lower degree and lymphoma remains the major cause of death of HIV patients. Most treatment procedures disclose a relatively poor outcome of patients with low response rates, high number of relapses and AIDS events. Since the majority of HIV-associated NHL are CD20-positive the addition of rituximab to the standard regimen - CHOP could improve the outcome of these patients

ELIGIBILITY:
Inclusion Criteria:

* HIV positive with a high grade Ann Arbor stage I to IV untreated non-Hodgkin's lymphoma of B-cell origin confirmed by biopsy. The following histologies are eligible: *Burkitt's lymphoma, *diffuse large B-cell with standard histological diagnosis, *Burkitt-like and high grade large cell immunoblastic lymphoma with immunophenotyping CD20 positive
* Good and intermediate prognostic group (no more than one of the following prognostic factors: *CD4 below 100/µl, *history of opportunistic infection, *Karnofsky index below 60 percent or ECOG over 2)
* Written inform consent to participate

Exclusion Criteria:

* Active viral hepatitis
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 1999-01; Study Completion 2003-10

PRIMARY OUTCOMES:
Evaluate the response rate of lymphoma treated

SECONDARY OUTCOMES:
Duration of response
Evaluate the time to progression
Survival
Safety of rituximab in HIV patients with lymphoma when sequentially administered with chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Francois Boue, MD, Principal Investigator — Service de Medecine Interne Hopital A Beclere Clamart France; Dominique Costagliola, Study Chair — Inserm U 720
Locations (1):
- Service de Medecine Interne Hopital Antoine Beclere, Clamart, France